CLINICAL TRIAL: NCT05150015
Title: ElastoMeric Infusion Pumps for Hospital AntibioTICs
Acronym: EMPHATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stuart Bond (Other)
Responsible Party: Sponsor-Investigator, Stuart Bond, Co-chief investigator, Mid Yorkshire Teaching NHS Trust
Organization: Mid Yorkshire Teaching NHS Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21/1358
Record Dates: First submitted 2021-11-22; First posted 2021-12-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Pilot feasability study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Number of consented patients who complete the antibiotics through an elastomeric pump (Experimental): Flucloxacillin, piperacillin/taozbactam and benzylpenicillin will be use
  Interventions: Device: To assess the feasibility of giving intravenous antibiotics to adult inpatients using elastomeric infusion pumps (EMPs)

INTERVENTIONS:
Device: To assess the feasibility of giving intravenous antibiotics to adult inpatients using elastomeric infusion pumps (EMPs) — Single arm study

SUMMARY:
Special pumps called self-deflating Elastomeric Pumps (EMPs) will be tested for giving antibiotics via a drip to hospital patients. EMPs are filled with antibiotics, attached to a "drip" (usually in the arm) and worn on the body, slowly giving antibiotics through the day. EMPs are often used to give antibiotics to patients in their own home but they have not been used to treat patients in hospital before, so a small study of 10 patients will be conducted to see if a full scale clinical trial is worthwhile. EMPs will be tested for ease of use and safety in hospital, and to find out what staff and patients think about them. The pilot will be done to see if a clinical trial would be good value for money by comparing time spent in hospital, nursing time and overall cost to the NHS of the two ways of giving antibiotics to patients.

DETAILED DESCRIPTION:
4 Background 4.1 Antibiotic resistance Antibiotic resistance (AMR) is when bacteria have changed (mutated) so they can survive the effects of antibiotics, meaning antibiotics are less effective. AMR is a major threat to health worldwide. In UK hospitals, at least a third of patients are on antibiotics at any given time. Hospital patients with serious infections are often given intravenous antibiotics (through a "drip" into a vein). Cutting down unnecessary antibiotic prescribing is key to reducing resistance.

4.2 Problems giving intravenous antibiotics Giving intravenous antibiotics takes a lot of nursing time. This is made worse if antibiotics are needed more than once a day. Nurses are the only staff who give intravenous antibiotics in hospitals, and there is a shortage of 40,000 nurses in the NHS. Because of this, it is common for doses to be missed. The COVID-19 pandemic has increased the pressure on nurses' time. It is not always practical to give antibiotics 4 or 6 times a day so less effective antibiotics may be used instead.

4.3 What can be done to help? Some antibiotics work better when given slowly into a vein all the time. EMPs are self-powered devices that deliver antibiotics in this way.

EMPs:

* are currently used to give antibiotics to patients in their own homes
* are not used to give antibiotics to patients in hospitals because the safety, benefits and value for money have not been confirmed
* could allow more nurse time for patient care by reducing the time to set up antibiotic drips.
* could make things better for patients by allowing them to move more, sleep better, recover faster and spend less time in hospital

4.4 Designs and methods used Patients who could have antibiotics through EMPs will be identified from clinical ward rounds. EMPs will be tested for safety in hospital patients, as well as value for money in the NHS by collecting information about costs, nursing time and length of hospital stay. Surveys of patients and nursing staff will be conducted to explore how EMPs could be best used in hospital.

4.5 Patient and public involvement (PPI) This research has been driven by patients who know how difficult it is to keep mobile when attached to drip stands; how disturbed sleep from drips being set up in the night affects their wellbeing; and, how they are concerned about missed doses of antibiotics. The project has been designed with input from a PPI representative (Co-investigator Thompson) who has reviewed all project plans and materials.

4.6 Dissemination Findings will be published in medical journals and presented at conferences/NHS patient events. Social media will be used to let people know what is found and infographics will be developed to help communicate findings using social media. If appropriate, funding will be sought for a full trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years and over admitted to hospital with an infection requiring treatment for 7 days or more with intravenous flucloxacillin, piperacillin/tazobactam or benzylpenicillin Clinically stable and improving as assessed by the hospital medical consultant and likely to be well enough for discharge in the next two weeks.

Able to provide written consent or witnessed consent

Exclusion Criteria:

* Unable to receive an appropriate vascular access device, such as a peripherally inserted central catheter (PICC) Penicillin allergy and unsuitable to receive penicillin challenge or desensitisation.

Requires a combination of intravenous antibiotics, any of which needs to be given more often than once daily.

Requires transfer to another hospital Unsuitable for outpatient parenteral antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Number (%) of consented inpatients who complete the planned course of intravenous antibiotics through an EMP | 6 months

SECONDARY OUTCOMES:
Number (%) of screened patients as identified by a microbiologist, antimicrobial pharmacist or the patient's clinical team | 6 months
Number (%) of screened patients consented (recruitment) | 6 months
Number (%) of consented patients who receive ≥1 dose of EMP | 6 months
Time (hrs) from electronic prescribing (with planned start date) of initial intravenous antibiotic to administration of first dose through EMP | 6 months
Time (hrs) from identification of medically fit for discharge to actual discharge | 6 months
Duration of hospital inpatient stay (days) | 6 months
Time (minutes) to order, procure, deliver and administer EMPs | 6 months
Clinical cure (resolution of symptoms) assessed by hospital medical consultant | 6 months
30-day mortality | 6 months
High residual volume in EMP (greater than 15% of 240mL = 36mL) | 6 months
Duration of total antibiotic course (days), including any early termination of planned treatment course and reason | 6 months
Description of antibiotic treatment pathway: intermittent, EMP, outpatient parenteral antibiotic therapy (OPAT), oral, cease | 6 months
Number of intravascular access devices required, including intermittent infusion period and EMP period | 6 months
Number (%) of missed and delayed doses from beginning of antibiotic course, either with intermittent infusion or EMP | 6 months
Time taken (hrs) to order, procure, deliver and administer antibiotics through EMPs | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mid Yorkshire Hospitals NHS Trust, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No